CLINICAL TRIAL: NCT07339098
Title: A Prospective, Multicenter, Single-arm, Open-label, Non-randomized Exploratory Clinical Trial to Evaluate the Efficacy and Safety of Glomerular Filtration Rate (GFR-EPI) Using NEFRONIX in Patients With Chronic Kidney Disease (CKD)
Brief Title: Efficacy and Safety of the Ultrasound Stimulation Device NEFRONIX in Patients With Chronic Kidney Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anasonic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cenovia; 1866 (Other: Ministry of Food and Drug Safety (MFDS))
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- NEFRONIX Treatment (Experimental): Participants in this arm will receive ultrasound stimulation using the NEFRONIX G-01 device applied to the kidneys three times per week for four weeks, in accordance with the study protocol. Standard clinical care for chronic kidney disease will be maintained throughout the study period.
  Interventions: Device: Ultrasound Stimulation (NEFRONIX G-01)

INTERVENTIONS:
Device: Ultrasound Stimulation (NEFRONIX G-01) — Ultrasound stimulation will be delivered to the renal area using the NEFRONIX G-01 device. The intervention will be administered three times per week for four weeks in accordance with the study protocol. Standard clinical management for chronic kidney disease will be continued during the study period.

SUMMARY:
This study is a prospective, multicenter, single-arm, open-label, non-randomized exploratory clinical trial designed to evaluate the safety and potential efficacy of an ultrasound stimulation device (NEFRONIX G-01) in patients with chronic kidney disease (CKD). Baseline functional assessments will be performed prior to intervention. Participants will receive ultrasound stimulation applied to the kidneys three times per week for four weeks according to the study protocol. Clinical evaluations will be conducted at baseline, at the end of treatment, and 12 weeks after completion of treatment. Renal function will be assessed using changes in estimated glomerular filtration rate based on serum creatinine (CKD-EPI eGFR Cr) and cystatin C (CKD-EPI eGFR CysC). Additional assessments will include imaging studies (Tc-99m DTPA renal scintigraphy and renal ultrasonography), urinalysis for proteinuria, inflammatory markers (high-sensitivity C-reactive protein), and renal injury biomarkers (neutrophil gelatinase-associated lipocalin).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have received sufficient explanation of the study and have voluntarily provided written informed consent.
* Male and female adults aged 18 to 65 years at the time of consent.
* Participants with chronic kidney disease, defined as an estimated glomerular filtration rate (eGFR) between 20 and 60 mL/min/1.73 m².
* Participants who agree to use and maintain appropriate contraception throughout the study period.

Exclusion Criteria:

* Participants currently enrolled in another clinical study with an ongoing follow-up period.
* Participants with heart failure.
* Participants who have undergone reperfusion therapy for cardiovascular disease within the past year.
* Participants with platelet or coagulation disorders, including those receiving antithrombotic therapy.
* Participants with acute or chronic urinary tract infection.
* Participants with polycystic kidneys.
* Participants with anatomical kidney abnormalities (e.g., solitary kidney, horseshoe kidney, polycystic kidney disease) as determined by the investigator.
* Participants with urinary tract obstruction.
* Participants who have received a kidney transplant.
* Participants with kidney or urinary tract stones.
* Participants who have experienced acute kidney injury or changes in CKD stage within the past 3 months.
* Participants with serum albumin <3.0 g/dL and either 24-hour proteinuria ≥3.0 g/day or random urine protein/creatinine ratio ≥3.0 mg/mg.
* Participants with uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg despite treatment with two or more antihypertensive medications).
* Participants with liver dysfunction.
* Participants receiving immunosuppressive therapy.
* Participants with body mass index (BMI) >35 kg/m² or body weight <40 kg.
* Participants with a history of severe illness, such as cancer or tuberculosis.
* Participants with contact dermatitis or other significant skin sensitivities.
* Participants with fever ≥40°C (104°F) measured via tympanic temperature.
* Participants deemed unsuitable for participation in the study by the investigator for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Glomerular Filtration Rate Estimated by Serum Creatinine (eGFR-EPI Cr) | Baseline to after 4 weeks of application of the investigational medical device
  The primary outcome is the change in glomerular filtration rate estimated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation based on serum creatinine (eGFR-EPI Cr) from baseline to after 4 weeks of application of the investigational medical device.

SECONDARY OUTCOMES:
Change in Glomerular Filtration Rate Estimated by Serum Creatinine (eGFR-EPI Cr) | Baseline to 12 weeks after application of the investigational medical device
Change in Glomerular Filtration Rate Estimated by Cystatin C (eGFR-EPI CysC) | Baseline to after 4 weeks of application of the investigational medical device
Change in Glomerular Filtration Rate Estimated by Cystatin C (eGFR-EPI CysC) | Baseline to 12 weeks after application of the investigational medical device
Change From Baseline in Urinary Protein Excretion | Baseline to after 4 weeks of application of the investigational medical device
Change From Baseline in Urinary Protein Excretion | Baseline to 12 weeks after application of the investigational medical device
Change From Baseline in Serum High-Sensitivity C-Reactive Protein (hsCRP) Concentration | Baseline to after 4 weeks of application of the investigational medical device
Change From Baseline in Serum High-Sensitivity C-Reactive Protein (hsCRP) Concentration | Baseline to 12 weeks after application of the investigational medical device
Change From Baseline in Renal Resistive Index Assessed by Doppler Ultrasonography | Baseline to after 4 weeks of application of the investigational medical device
Change From Baseline in Renal Resistive Index Assessed by Doppler Ultrasonography | Baseline to 12 weeks after application of the investigational medical device
Change From Baseline in Serum Neutrophil Gelatinase-Associated Lipocalin (NGAL) Concentration | Baseline to after 4 weeks of application of the investigational medical device
Change From Baseline in Serum Neutrophil Gelatinase-Associated Lipocalin (NGAL) Concentration | Baseline to 12 weeks after application of the investigational medical device
Change in Renal Function Assessed by Tc-99m DTPA Renal Scintigraphy | Baseline to after 4 weeks of application of the investigational medical device
Change in Renal Function Assessed by Tc-99m DTPA Renal Scintigraphy | Baseline to 12 weeks after application of the investigational medical device

IPD SHARING:
Plan to Share IPD: No